CLINICAL TRIAL: NCT02876575
Title: A Prospective, Multi-center, Single Arm Non-comparative Pilot Study of BiZact™ on Adults Undergoing Tonsillectomy
Brief Title: A Study of BiZact™ on Adults Undergoing Tonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVBZTS0562
Record Dates: First submitted 2016-07-29; First posted 2016-08-24 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Tonsillectomy
MeSH Terms: interventions — Tonsillectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- A bipolar instrument for tonsillectomies (Other): A bipolar electrosurgical device that employs RF energy and pressure to ligate vessels interposed between its jaws which can then be transected using the built in knife deployed by the device trigger.
  Interventions: Device: A bipolar instrument for tonsillectomies

INTERVENTIONS:
Device: A bipolar instrument for tonsillectomies — A bipolar electrosurgical device that employs RF energy and pressure to ligate vessels interposed between its jaws which can then be transected using the built in knife deployed by the device trigger.

SUMMARY:
The purpose of this study is to assess the severity of post-operative pain following the use of the BiZact™ device in adult (≥22 years of age in United States and ≥18 years of age in Europe) tonsillectomy procedures.

DETAILED DESCRIPTION:
Study Design: Prospective, multi-center, single-arm non-comparative pilot study to assess the severity of post-operative pain with the use of BiZact™ for tonsillectomy.

Study Visits:

* Screening
* Surgery, Day 0
* Post-Op Follow-up Day 1 - Day 7 & Day 10 (Home assessments)
* Post-Op Follow-up Day 14 (Office Visit)

ELIGIBILITY:
Inclusion Criteria:

1. Adults (male or female) ≥22 in United States and ≥18 years of age in Europe years of age
2. Scheduled to undergo tonsillectomy
3. Signed informed consent by subject

Exclusion Criteria:

1. Subjects undergoing:

   1. Simultaneous adenoidectomy
   2. Tonsillectomy as a result of cancer
   3. Unilateral tonsillectomy
   4. Current participation in other clinical trials
2. Subjects with:

   1. Current tobacco use
   2. Known bleeding disorders
   3. History of peritonsillar abscess
   4. Craniofacial disorders
   5. Down syndrome (Trisomy 21)
   6. Cerebral palsy
   7. Major heart disease (including but not limited to; right-sided heart failure, left-sided heart failure, congestive heart failure, coronary artery disease, arrhythmias, chronic heart failure, acute heart failure, etc.)
   8. Subjects unable to comply with the required study follow-up visits
   9. Pregnancy
3. The subject has comorbidities which, in the opinion of the investigator, will not be appropriate for the study or the subject has an estimated life expectancy of less than 6 months
4. Any subject who is considered to be part of a vulnerable population (e.g. prisoners or those without sufficient mental capacity)
5. The subject has participated in any drug or device research study within 30 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Karni, MD, Principal Investigator — University of Texas at Houston
Locations (2):
- UT Health, Houston, Texas, United States
- Sophia Hemmet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 48 Adults, greater than or equal to 22 in the US and greater than or equal to 18 in Europe, were enrolled into a single-arm trial. A total of 50 subjects were screened and consented and 2 subjects were withdrawn due to physician request.
Groups:
- BiZact Arm: A bipolar electrosurgical device that employs RF energy and pressure to ligate vessels interposed between its jaws which can then be transected using the built in knife deployed by the device trigger.
Period: Overall Study
Arm/Group | BiZact Arm
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adults (male or female) ≥22 years of age in United States and
  ≥18 years of age in Europe 2. Scheduled to undergo tonsillectomy 3. Signed informed consent by subject
Groups:
- BiZact Arm: 48 adults undergoing tonsillectomy
Arm/Group | BiZact Arm
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 46
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 24
  United States | 26
Undergoing Tonsillectomy [Count of Participants; unit: Participants] | 48
Signed Informed Consent [Count of Participants; unit: Participants] | 48

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessment Using a Visual Analog Scale (VAS)
Description: The severity of post-operative pain following the use of the BiZact™ device in adult (≥22 years of age in United States and ≥18 years of age in Europe) tonsillectomy procedures will be analyzed at each post-operative assessment: at days 1 through 7, 10 and 14. This pain score will be assessed quantitatively using the VAS scale and qualitatively using the below subgroups:
  * No Pain: VAS= 0
  * Mild Pain: VAS > 0 and < 4
  * Moderate: VAS ≥ 4 and < 7
  * Severe: VAS ≥ 7
Time Frame: Post-operative Day 1
Population: 46 out of 48 subjects completed the post-operative assessment as directed by the protocol, 2 subjects did not completed the assessment on day 1 as directed by the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 46
units on a scale | 5.4 (2.59)

2. Primary Outcome: Pain Assessment Using a Visual Analog Scale (VAS)
Description: as for outcome 1
Time Frame: Post-operative Day 2
Population: 46 out of 48 subjects completed the post-operative assessment as directed by the protocol, 2 subjects did not completed the assessment on day 2 as directed by the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 46
units on a scale | 5.9 (2.36)

3. Primary Outcome: Pain Assessment Using a Visual Analog Scale (VAS)
Description: as for outcome 1
Time Frame: Post-operative Day 3
Population: 45 out of 48 subjects completed the post-operative assessment as directed by the protocol, 3 subjects did not completed the assessment on day 3 as directed by the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 45
units on a scale | 6.1 (2.05)

4. Primary Outcome: Pain Assessment Using a Visual Analog Scale (VAS)
Description: as for outcome 1
Time Frame: Post-operative Day 4
Population: 46 out of 48 subjects completed the post-operative assessment as directed by the protocol, 2 subjects did not completed the assessment on day 4 as directed by the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 46
units on a scale | 6.3 (2.01)

5. Primary Outcome: Pain Assessment Using a Visual Analog Scale (VAS)
Description: as for outcome 1
Time Frame: Post-operative Day 5
Population: 46 out of 48 subjects completed the post-operative assessment as directed by the protocol, 2 subjects did not completed the assessment on day 5 as directed by the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 46
units on a scale | 6.3 (2.16)

6. Primary Outcome: Pain Assessment Using a Visual Analog Scale (VAS)
Description: as for outcome 1
Time Frame: Post-operative Day 6
Population: 46 out of 48 subjects completed the post-operative assessment as directed by the protocol, 2 subjects did not completed the assessment on day 6 as directed by the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 46
units on a scale | 6.0 (2.25)

7. Primary Outcome: Pain Assessment Using a Visual Analog Scale (VAS)
Description: as for outcome 1
Time Frame: Post-operative Day 7
Population: 46 out of 48 subjects completed the post-operative assessment as directed by the protocol, 2 subjects did not completed the assessment on day 7 as directed by the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 46
units on a scale | 4.9 (2.54)

8. Primary Outcome: Pain Assessment Using a Visual Analog Scale (VAS)
Description: as for outcome 1
Time Frame: Post-operative Day 10
Population: 46 out of 48 subjects completed the post-operative assessment as directed by the protocol, 2 subjects did not completed the assessment on day 10 as directed by the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 46
units on a scale | 2.7 (2.54)

9. Primary Outcome: Pain Assessment Using a Visual Analog Scale (VAS)
Description: as for outcome 1
Time Frame: Post-operative Day 14
Population: 46 out of 48 subjects completed the post-operative assessment as directed by the protocol, 2 subjects did not completed the assessment on day 14 as directed by the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 46
units on a scale | 1.2 (1.78)

10. Secondary Outcome: Time to Normal Diet Following the Use of the BiZact™ Device in Adult (≥22 Years of Age in United States and ≥18 Years of Age in Europe) Tonsillectomy Procedures
Description: Ability to return to Normal, subject's baseline, diet. EORTC Quality of Life Questionnaire (EORTC QLQ -H&N35) will be analyzed at each post-operative assessment: at days 1 through 7, 10 and 14. The module consists of 35 questions assessing symptoms and side effects of treatment, social function, and body image/sexuality. The head and neck cancer module incorporates seven multi-item scales that assess pain, swallowing, senses (taste and smell), speech, social eating, social contact, and sexuality. There are also eleven single items. For all items and scales, high scores indicate more problems. This score will be assessed qualitatively by asking if they have experienced symptoms or problems using the below subgroups:
  * Not at all: 1
  * A little: 2
  * Quite a bit: 3
  * Very much: 4
Time Frame: Post-operative Day 28
Measure: Mean (Standard Deviation); unit: days
Arm/Group | BiZact Arm
Number analyzed (Participants) | 48
days | 12.3 (2.57)

11. Secondary Outcome: Time to Normal Activity Following the Use of the BiZact™ Device in Adult (≥22 Years of Age in United States and ≥18 Years of Age in Europe) Tonsillectomy Procedures
Description: Ability to return to Normal, subject's baseline, activity. EORTC Quality of Life Questionnaire (EORTC QLQ -H&N35) will be analyzed at each post-operative assessment: at days 1 through 7, 10 and 14. The module consists of 35 questions assessing symptoms and side effects of treatment, social function, and body image/sexuality. The head and neck cancer module incorporates seven multi-item scales that assess pain, swallowing, senses (taste and smell), speech, social eating, social contact, and sexuality. There are also eleven single items. For all items and scales, high scores indicate more problems. This score will be assessed qualitatively by asking if they have experienced symptoms or problems using the below subgroups:
  * Not at all: 1
  * A little: 2
  * Quite a bit: 3
  * Very much: 4
Time Frame: Post-operative Day 28
Measure: Mean (Standard Deviation); unit: days
Arm/Group | BiZact Arm
Number analyzed (Participants) | 48
days | 12.4 (2.77)

ADVERSE EVENTS:
Time Frame: Adverse Events were collects from baseline and day 0 to 14 days follow up
Description: In alignment with ISO 14155:2011 (Section 3.2), an Adverse Event is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device. This definition includes events related to the investigational medical device and the procedures involved.
Arm/Group | BiZact Arm
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 6/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BiZact Arm (N=48)
Post-Tonsillectomy Hemorrhage (Injury, poisoning and procedural complications) | 5 (6)
Pain (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Medical Center /Investigator may publish the results of work performed under this Agreement, in accordance with the Publication Policy described in the Clinical Investigation Plan and publication guidelines from the Declaration of Helsinki; provided, however, that any such Publication shall be at a time determined by Medtronic and shall be provided to Medtronic for review at least sixty (60) days prior to submission or presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT02876575/Prot_SAP_000.pdf